CLINICAL TRIAL: NCT00325156
Title: An Open, Multicentric, Post-marketing Surveillance Study to Assess the Safety and Reactogenicity of GlaxoSmithKline Biologicals' DTPa-IPV/Hib Vaccine Administered at 3, 4, 5 and 18 Months of Age, in Healthy Infants.
Brief Title: Assess the Safety & Reactogenicity of DTPa-IPV/Hib Vaccine Administered at 3, 4, 5 & 18 Mths of Age, in Healthy Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 100917; 2015-001512-35 (EudraCT Number)
Record Dates: First submitted 2006-02-08; First posted 2006-05-12 (Estimated); Results first posted 2017-02-07 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Diphtheria; Tetanus; Poliomyelitis; Acellular Pertussis; Haemophilus Influenzae Type b; Diphtheria-Tetanus-aPertussis-Poliomyelitis Vaccines
MeSH Terms: conditions — Diphtheria; Tetanus; Poliomyelitis; Haemophilus Infections

ARMS (1):
- Group A (Experimental)
  Interventions: Biological: GSK Biologicals' combined DTPa-IPV/Hib vaccine

INTERVENTIONS:
Biological: GSK Biologicals' combined DTPa-IPV/Hib vaccine — 4 intramuscular injections

SUMMARY:
To assess the safety and reactogenicity of the DTPa-IPV/Hib vaccine as primary and booster vaccination. The DTPa-IPV/Hib vaccine given at 3 and 4 months of age is co-administered with GSK Biologicals' rotavirus vaccine or Placebo.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
Single group study. Subjects in GSK Biologicals' rotavirus study (Rota-028) in Singapore will be enrolled in this study. 3-4-5 month schedule with a booster dose at 18 months

ELIGIBILITY:
Inclusion criteria

* Subjects must have been enrolled in the Rota-028 study.
* A male or female between, and including, 11 and 17 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol

Exclusion criteria

* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs during the study period.
* Planned administration/ administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of the vaccine and ending 30 days after.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.

Ages: 11 Weeks to 17 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2590 (Actual)
Dates: Start 2004-11-02 (Actual); Primary Completion 2007-08-23 (Actual); Study Completion 2007-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=350

REFERENCES:
- [Background] Lim FS, Phua KB, Lee BW, Quak SH, Teoh YL, Ramakrishnan G, Han HH, Van Der Meeren O, Jacquets JM, Bock HL. Safety and reactogenicity of DTPa-HBV-IPV/Hib and DTPa-IPV/I-Hib vaccines in a post-marketing surveillance setting. Southeast Asian J Trop Med Public Health. 2011 Jan;42(1):138-47. PMID 21323176
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 100917 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 100917 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 100917 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 100917 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 100917 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 100917 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Infanrix-IPV+Hib Group: Healthy male or female subjects between and including 11 to 17 weeks of age at the time of first vaccination, who previously participated in a human rotavirus (HRV) study (444563/028), received 3 primary doses and one booster dose of Infanrix™-IPV/Hib vaccine at 3,4 and 5 months of age and 18 months of age, respectively, administered intramuscularly into the anterolateral thigh. Subjects also received 2 oral doses of Rotarix™ (HRV) vaccine or placebo, at 3 and 4 months of age.
Period: Overall Study
Arm/Group | Infanrix-IPV+Hib Group
Started | 2590
Completed | 2478
Not Completed | 112
Not completed — Protocol Violation | 8
Not completed — Lost to follow-up (complete vaccination) | 41
Not completed — Migrated/moved from study area | 12
Not completed — Adverse event, non-fatal | 3
Not completed — Lost to follow-up (incompl. vaccination) | 16
Not completed — Other | 1
Not completed — Withdrawal by Subject | 31

BASELINE CHARACTERISTICS:
Groups:
- Infanrix-IPV+ Hib Group: Healthy male or female subjects between and including 11 to 17 weeks of age at the time of first vaccination, who previously participated in a human rotavirus (HRV) study (444563/028), received 3 primary doses and one booster dose of Infanrix™-IPV/Hib vaccine at 3,4 and 5 months of age and 18 months of age, respectively, administered intramuscularly into the anterolateral thigh. Subjects also received 2 oral doses of Rotarix™ (HRV) vaccine or placebo, at 3 and 4 months of age.
Arm/Group | Infanrix-IPV+ Hib Group
Number analyzed (Participants) | 2590
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 13.3 (0.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1245
  Male | 1345

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any Solicited Local and General Symptoms
Description: Assessed solicited local and general symptoms were pain, redness, swelling, drowsiness, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C )], irritability and loss of appetite. Any was defined as any report of the specified symptom irrespective of intensity grade and relationship to vaccination.
Time Frame: During the 4-day (Days 0-3) post-vaccination period, across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and who had filled-in the symptom sheet.
Measure: Number; unit: Subjects
Arm/Group | Infanrix-IPV+Hib Group
Number analyzed (Participants) | 2580
Subjects
  Any Pain, Across doses | 855
  Any Redness, Across doses | 907
  Any Swelling, Across doses | 706
  Any Drowsiness, Across doses | 929
  Any Fever (Axillary/≥ 37.5°C), Across doses | 1482
  Any Irritability, Across doses | 1217
  Any Loss of appetite, Across doses | 1010

2. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 30-day (Days 0-29) post-vaccination period
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Number; unit: Subjects
Arm/Group | Infanrix-IPV+Hib Group
Number analyzed (Participants) | 2590
Subjects | 914

3. Secondary Outcome: Number of Subjects Reporting Large Injection Site Swelling
Description: A large swelling reaction was defined as swelling with a diameter greater than (>) 50 millimeters (mm), noticeable diffuse swelling or noticeable increase of limb circumference.
Time Frame: At Month 18, post-booster dose
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Infanrix-IPV+Hib Group
Number analyzed (Participants) | 2540
Subjects
  Local swelling | 10
  Diffuse swelling | 1

4. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Infanrix-IPV+Hib Group
Number analyzed (Participants) | 2590
Subjects | 380

ADVERSE EVENTS:
Time Frame: Solicited local and general adverse events (AEs): during the 4-day (Days 0-3) after vaccination. Unsolicited local and general AEs: during the 30-day (Days 0-29) after vaccination. Serious adverse events (SAEs): during the entire study period.
Arm/Group | Infanrix-IPV+Hib Group
Serious Adverse Events (participants affected / at risk) | 380/2590
Other Adverse Events (participants affected / at risk) | 2167/2590
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix-IPV+Hib Group (N=2590)
Kawasaki's disease (Vascular disorders) | 6
Haematoma (Vascular disorders) | 2
Milk allergy (Immune system disorders) | 1
Pyrexia (General disorders) | 1
Swelling (General disorders) | 1
Balanitis (Reproductive system and breast disorders) | 2
Head injury (Injury, poisoning and procedural complications) | 12
Foreign body trauma (Injury, poisoning and procedural complications) | 3
Thermal burn (Injury, poisoning and procedural complications) | 3
Arthropod bite (Injury, poisoning and procedural complications) | 2
Skin laceration (Injury, poisoning and procedural complications) | 2
Accidental exposure (Injury, poisoning and procedural complications) | 1
Burns second degree (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Skull fracture (Injury, poisoning and procedural complications) | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Cardiac aneurysm (Cardiac disorders) | 1
Cryptorchism (Congenital, familial and genetic disorders) | 1
Laryngomalacia (Congenital, familial and genetic disorders) | 1
Lymphangioma (Congenital, familial and genetic disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 11
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Febrile convulsion (Nervous system disorders) | 25
Convulsion (Nervous system disorders) | 7
Benign intracranial hypertension (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Gastritis (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 3
Intussusception (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Vesicoureteric reflux (Renal and urinary disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 3
Petechiae (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Urticaria chronic (Skin and subcutaneous tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Failure to thrive (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Bronchiolitis (Infections and infestations) | 87
Upper respiratory tract infection (Infections and infestations) | 47
Gastroenteritis (Infections and infestations) | 45
Bronchitis (Infections and infestations) | 20
Gastritis viral (Infections and infestations) | 16
Urinary tract infection (Infections and infestations) | 16
Escherichia urinary tract infection (Infections and infestations) | 13
Hand-foot-and-mouth disease (Infections and infestations) | 13
Viral infection (Infections and infestations) | 13
Gastroenteritis viral (Infections and infestations) | 12
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 10
Gastroenteritis rotavirus (Infections and infestations) | 7
Herpangina (Infections and infestations) | 7
Pneumonia (Infections and infestations) | 7
Abscess limb (Infections and infestations) | 6
Pharyngitis (Infections and infestations) | 6
Viral upper respiratory tract infection (Infections and infestations) | 6
Gastroenteritis salmonella (Infections and infestations) | 5
Lobar pneumonia (Infections and infestations) | 4
Lower respiratory tract infection (Infections and infestations) | 4
Viral skin infection (Infections and infestations) | 4
Subcutaneous abscess (Infections and infestations) | 3
Bronchopneumonia (Infections and infestations) | 2
Croup infectious (Infections and infestations) | 2
Haematoma infection (Infections and infestations) | 2
Otitis media (Infections and infestations) | 2
Perianal abscess (Infections and infestations) | 2
Abscess (Infections and infestations) | 1
Acarodermatitis (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Conjunctivitis viral (Infections and infestations) | 1
Dengue fever (Infections and infestations) | 1
Epstein-barr virus infection (Infections and infestations) | 1
Exanthema subitum (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastroenteritis bacterial (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Lymphadenitis bacterial (Infections and infestations) | 1
Necrotising fasciitis (Infections and infestations) | 1
Parainfluenzae viral laryngotracheobronchitis (Infections and infestations) | 1
Parotitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Viral pharyngitis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix-IPV+Hib Group (N=2590)
Cough (Respiratory, thoracic and mediastinal disorders) | 146
Pain (General disorders) | 855
Redness (General disorders) | 907
Swelling (General disorders) | 706
Drowsiness (General disorders) | 929
Fever (Axillary) (General disorders) | 1482
Irritability (General disorders) | 1217
Loss of appetite (General disorders) | 1010
Upper respiratory tract infection (Infections and infestations) | 391

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.